CLINICAL TRIAL: NCT04002869
Title: Innovation in Tuberculosis
Acronym: INNOVA4TB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut Germans Trias i Pujol (Other)
Collaborators: Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government); Umeå University (Other); North-Western State Medical University named after I.I.Mechnikov (Other); INSTITUTUL DE FTIZIOPNEUMOLOGIE CHIRIL DRAGANIUC (Unknown); ODESA SIGNIFICANT DISEASES CENTER (Unknown); Vinnitsa National Medical University (Other); SERVICIOS CLINICOS SA (Unknown); Genome Identification Diagnostics GmbH (Unknown); EMPE DIAGNOSTICS AB (Unknown); MAGRITEK GMBH (Unknown); Universidad de La Frontera (Other)
Responsible Party: Principal Investigator, Jose Antonio Dominguez Benitez, Senior Researcher, Fundació Institut Germans Trias i Pujol
Other Study IDs: 823854
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Active TB suspicion: This study will include both adults and children with suspicion of different degrees of severity of active TB (pulmonary and extrapulmonary) to bring the investigator's study population into line with the routine clinical practice and to avoid the spectrum bias
  Interventions: Diagnostic Test: Immunologic, molecular, metabolomic and radiolologic diagnostic
- Latent TB infection: Individuals with latent TB infection (adults and children), with positive TST and/or IGRAs; without any sign or radiological evidence of TB disease or any clinical picture compatible with the criteria defined in the section TB cases.
  Interventions: Diagnostic Test: Immunologic, molecular, metabolomic and radiolologic diagnostic
- NTM infection: Adult and pediatric patients with lymphadenopathies caused by NTMs or individuals with chronic respiratory diseases with a NTM microbiologically confirmed by culture isolation.
  Interventions: Diagnostic Test: Immunologic, molecular, metabolomic and radiolologic diagnostic
- Uninfected control: Both adult and children without active TB and no immunologic evidence of M. tuberculosis infection, with negative TST and/or IGRAs
  Interventions: Diagnostic Test: Immunologic, molecular, metabolomic and radiolologic diagnostic
- Other respiratory diseases: Subjects with ARIs, and subjects with lung cancer; without any clinical picture compatible with the criteria defined in TB cases section. Patients with ARIs will be identified as individuals with clinical signs, symptoms and radiology of respiratory infections, and microbiological confirmation of non-TB origin. Patients with lung cancer will be identified as those with a high clinical suspicion, a suggestive chest X-ray/computed tomography scan, and a confirmed histopathological/cytological diagnosis
  Interventions: Diagnostic Test: Immunologic, molecular, metabolomic and radiolologic diagnostic

INTERVENTIONS:
Diagnostic Test: Immunologic, molecular, metabolomic and radiolologic diagnostic — Evaluation and development of new technologies

SUMMARY:
Tuberculosis (TB) is one of the major infectious diseases worldwide, and the emergence and spread of drug resistant cases is a public health threat. However, the conventional methods used for diagnosis and drug-susceptibility testing are not enough for controlling the disease. In addition, all TB patients, independently of their age, gender, severity of the disease and type of responsible strain, follow the same treatment duration (up to 20 months in drug resistant cases), which often leads to high frequency of adverse events, suboptimal adherence to treatment, and poor outcome. Therefore, a transition from programmatic to personalized management of TB is needed.

INNOVA4TB proposal will develop innovative technologies and approaches in order to improve the individual risk assessment for TB development, to rapidly diagnose active TB, to detect the drug susceptibility of the strain, to design tailor-made therapies, and to use biomarkers to guide and individualize the duration of antimicrobial therapy. This is of great importance for improving the quality of life of patients and ensuring treatment success, as well as for economic reasons for the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* Immunosuppression will not be considered an exclusion criterion

Exclusion Criteria:

* Patients who are not able to give their informed consent to participate in the study will be excluded

Ages: 1 Month to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Briefly, subjects from different study groups will be included: (i) patients with suspicion of active TB, (ii) individuals with latent TB infection, (iii) patients with NTM infection, (iv) healthy uninfected controls, and (v) patients with other respiratory diseases such as Acute Respiratory Infections (ARIs) or lung cancer.
Sampling Method: Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | 01/01/2019 to 31/12/2022
  Sensitivity, Specificity and predictive values

CONTACTS AND LOCATIONS:
Locations (1):
- Institut D'Investigació Germans Trias I Pujol, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
the only possibility of sharing data it will be as anonymized data